CLINICAL TRIAL: NCT06728293
Title: Effect of the HCC Liver-Link Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lauren Nephew, Assistant Professor | Division of Gastroenterology & Hepatology| IU School of Medicine |IU Health Associate Vice Chair of Health Equity| IU School of Medicine | IU Health, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23696; 5K23MD018090 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-12-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: HCC; Racial Disparities

STUDY DESIGN:
Intervention Model Description: 20 patients will then be randomized to SOC and 20 to the Liver-Link Intervention. Randomization will be stratified by race and SES.
Masking Description: Participants will be randomized on a 1:1 basis, stratified by race and SES. NIH randomization tool will be used to randomize patients into status of care and intervention arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liver-Link Arm (Experimental): Those randomized to the Liver-Link portion of the study will proceed through the Liver-Link component intervention. Participation in this study will last 6 months. Participants in this group are assessed for knowledge of their disease, quality of life, substance use, and for social needs at the beginning of the program. Those who screen positive for social needs or high-risk alcohol will see social work. Participants will attend 3 support groups and compelte exit surveys. Participants will have 3 milestone checks during the 6 month study period and will be referred back to social work if they do not meet milestones. Participants will also have a knowledge assessment after a total of 2 HCC-related visits.
  Interventions: Other: Liver Link
- Standard of Care Arm (No Intervention): Individuals in the standard of care portion of the study will complete several questionnaires at the enrollment visit . Over the duration of study participation (6 months), participants in this arm may meet with a social worker as part of their standard health care treatment and will receive education via these standard of care visits. After at least two visits related to HCC clinical care, and participants in this arm will be contacted and will be asked to complete the knowledge assessment tool. At tne end of study they will complete exit survieys via redcap or phone.

INTERVENTIONS:
Other: Liver Link — Support Program
  Arms: Liver-Link Arm

SUMMARY:
This study is a pilot, multi-center randomized controlled trial testing the HCC Liver-Link intervention, a culturally tailored, multi-level program designed to reduce racial disparities in hepatocellular carcinoma (HCC) care. The intervention combines: (1) patient education to improve HCC-related disease and treatment knowledge, (2) social needs and substance use screening with referral to social work and community resources, and (3) facilitated access to subspecialty cancer care through a multidisciplinary HCC tumor board.

A total of 40 Black patients with Barcelona Clinic Liver Cancer (BCLC) stage 0, A, or downstaged B disease will be randomized to receive either the HCC Liver-Link intervention or usual care and followed for 6 months or until liver transplant waitlisting. Primary outcomes are time to receipt of curative therapies (liver transplantation or resection) and change in HCC-related knowledge. Findings will inform development of larger interventions to eliminate racial disparities in HCC outcomes.

ELIGIBILITY:
Inclusion Criteria

• Within UCSF criteria:

Candidates are eligible or a standardized MELD or PELD exception if, before completing locoregional therapy, they have lesions that meet one of the following criteria:

* One Class 5 lesion greater than 5 cm and less than or equal to 8 cm
* two or three Class 5 lesions that meeting all of the following

  * At least one lesion greater than 3cm
  * Each lesion less than or equal to 5 cm, and
  * A total diameter of all lesions less than or equal to 8cm
* Four or five Class 5 lesions each less than 3 cm, and a total diameter of all lesions less than or equal to 8 cm.
* Between 18-75 years old
* Have no more than two visits with an HCC-related provider
* Able to read, write, and speak English
* Any 1 of the following:

  * Self-report as Black race (can be multiple races as long as 1 is Black)
  * Self-report as insured by Medicaid (+/- Medicare)
  * SVI (Social vulnerability index) >= .75
  * Unmarried

Exclusion Criteria

* Lacks capacity to provide informed consent, including those with stage 2 HE or higher at the time of consent.
* Age over 75
* Last transthoracic echocardiogram with EF<40% (OK if no prior echo)
* BMI over 50
* Patients who, in the investigator's judgment, are unlikely to ever be eligible for liver transplantation or resection at the time of enrollment, with reason documented
* Prior history of any solid organ transplant
* Non-skin cancer malignancies other than hepatocellular carcinoma in past 2 years unless approved by PI (i.e. cervical cancer, early prostate cancer)
* Patients who have undergone resection or waitlisted
* Patients near completion of transplant evaluation, PI to determine utility of intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to waitlist | Up to 6 months post-enrollment
  Days from study enrollment to liver transplant waitlisting, assessed using OTTR.
Time to resection | Up to 6 months post-enrollment
  Days from study enrollment to surgical resection, assessed using EMR.
Waitlisting or Resection | Up to 6 months post-enrollment
  Proportion of participants who achieve liver transplant waitlisting or surgical resection, assessed using EMR and OTTR
Time to Death | Up to 12 months post-enrollment.
  Days from study enrollment to death, assessed using EMR and OTTR.

SECONDARY OUTCOMES:
HCC-Related Knowledge | Baseline and 6 months post-enrollment.
  Score on a 10-item internally developed HCC knowledge multiple-choice test.
Medical Mistrust | Baseline and 6 months post-enrollment.
  Score on 7-item Medical Mistrust Index.
Social Needs and AUD Linkage | Up to 6 months post-enrollment.
  Percentage of participants offered services for a social need, achieving improvement in a social need, and without alcohol use in the past 90 days; assessed by patient and social worker reports in REDCap.
Quality of Life (QOL) | Baseline and 6 months post-enrollment.
  Composite and domain-specific scores (anxiety, depression, social role participation) on PROMIS-29 QOL Tool.

OTHER OUTCOMES:
Feasibility | Ongoing through 6 months post-enrollment.
  Consent rate, reasons for decline, and percentage of visit completion (enrollment, support, social work), assessed in REDCap.
Usability | 6 months post-enrollment.
  Score on the Modified System Usability Scale assessing intervention binder.
Satisfaction | 6 months post-enrollment.
  Score on the Client Satisfaction Questionnaire (CSQ-8; range 25-100).
Fidelity | 6 months post-enrollment
  Percentage of scripted social support group content delivered across sites, assessed via transcript comparison.
Intervention Feedback - Patients | 6 months post-enrollment.
  Open-ended survey of patient satisfaction with support group content, binder content, and social work.
Intervention Feedback - Providers | 6 months post-enrollment.
  Open-ended survey assessing provider satisfaction with patient study participation and implementation of recommendations regarding social needs.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided